CLINICAL TRIAL: NCT06251271
Title: Diagnosing Obstructive Lung Disease With Point of Care Ultrasound- A Cross-sectional, Diagnostic Accuracy Test
Brief Title: Diagnosing Obstructive Lung Disease With Point of Care Ultrasound
Status: Completed | Type: Observational
Sponsor: Soroka University Medical Center (Other)
Collaborators: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Lior Fuchs MD, MD, Soroka University Medical Center
Other Study IDs: Protocol SOR-0185-23-CTIL; SCRC23032 (Other: Soroka Clinical Research Center); MOH_2023-10-04_012986 (Registry Identifier: Ministry of Health MyTrial)
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive; Asthma; COPD
Keywords: Point-of-Care Ultrasound; Dyspnea; Pulmonary Function Tests
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive; Asthma; Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Soroka University Medical Center Pulmonology Ward - 'All Comers': In the Pulmonology Ward, the cohort will encompass 'All Comers'-any patient referred for PFTs who meets the inclusion criteria. This cross-sectional observational study will screen all eligible patients presenting at the ward, offering a comprehensive snapshot of the diagnostic accuracy of point-of-care ultrasound in this diverse patient population.
  Interventions: Device: Point-of-Care Ultrasound
- Rabin Medical Center Pulmonology Ward - 'All Comers': In the Pulmonology Ward, the cohort will encompass 'All Comers'-any patient referred for PFTs who meets the inclusion criteria. This cross-sectional observational study will screen all eligible patients presenting at the ward, offering a comprehensive snapshot of the diagnostic accuracy of point-of-care ultrasound in this diverse patient population.
  Interventions: Device: Point-of-Care Ultrasound

INTERVENTIONS:
Device: Point-of-Care Ultrasound — Patients will undergo routine point-of-care ultrasound scans as part of the diagnostic process. The collected sonographic data and PFT results will assess point-of-care ultrasound's accuracy in diagnosing OLDs within the natural clinical setting.

SUMMARY:
The objective of this study is to evaluate the diagnostic accuracy of Point of Care Ultrasound (POCUS) in identifying obstructive lung diseases (OLDs), using pulmonary function tests (PFTs) as the gold standard for comparison.

DETAILED DESCRIPTION:
In this cross-sectional diagnostic accuracy test, 200 patients meeting the inclusion criteria will be enrolled to undergo random POCUS scans at the respiratory institute of Soroka University Medical Center. These patients, referred for PFTs, will be provided with a sonographic score based on several criteria. The study aims to capture comprehensive data, including sonographic results and medical history, to assess the sensitivity, specificity, PPV, and NPV of POCUS in diagnosing OLDs. Data management and analysis will be the responsibility of the Soroka Clinical Research Center, ensuring rigorous oversight and reliable results.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above
* Referral for full pulmonary function tests (PFTs)
* Patients are willing and able to sign a written informed consent form.

Exclusion Criteria:

* Unable to give written informed consent.
* Unable to remain supine.
* Poor effort at PFTs
* Subcutaneous emphysema

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will be screened at the respiratory institute of Soroka University Medical Center and will include patients who are referred for pulmonary function tests (PFTs) for any reason.
Sampling Method: Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-27 (Actual)

PRIMARY OUTCOMES:
Title: Comparative Accuracy of Point-of-Care Ultrasound and Pulmonary Function Tests in Respiratory Assessment | 12 Months
  This study aims to develop and validate a sonographic scoring system for Point-of-Care Ultrasound (POCUS) exams, using a scale from 0 to 10, where higher scores indicate worse respiratory function. The accuracy of POCUS in assessing respiratory function will be directly compared with outcomes from Pulmonary Function Tests (PFTs). Outcome measures will include the sensitivity, specificity, and overall accuracy of the sonographic scoring system in detecting respiratory abnormalities, alongside a comparison of diagnostic agreement between POCUS exams and PFT results.

SECONDARY OUTCOMES:
Correlation Between Sonographic Score and CT Scan Results | 12 Months
  This outcome will measure the correlation coefficient between the sonographic scoring system (scale of 0 to 10, with higher scores indicating worse outcomes) and CT scan results in detecting respiratory abnormalities. The aim is to quantify the strength and direction of the association between sonographic scores and objective findings on CT scans.
Sonographic Score Relationship with mMRC Dyspnea Scale | 12 Months
  This outcome will report the correlation between sonographic scores (on a scale of 0 to 10, where higher scores signify worse respiratory function) and the modified Medical Research Council (mMRC) dyspnea scale scores. The mMRC scale, ranging from 0 (no dyspnea) to 4 (severe dyspnea), assesses the severity of dyspnea. The analysis will measure how variations in sonographic scores align with patient-reported severity of dyspnea.
Sonographic Score Correlation with Diffusion Lung Capacity (DLCO) | 12 Months
  The objective is to measure the correlation between sonographic scores (scale of 0 to 10, with higher scores indicating worse respiratory status) and diffusion lung capacity (DLCO) values. This outcome will report the strength of association between sonographic findings and DLCO measurements, providing insights into respiratory function.
Sonographic Predictors of Obstructive Lung Disease Diagnosis | 12 Months
  This outcome will identify and quantify the predictive value of specific sonographic components for the diagnosis of Obstructive Lung Disease (OLD), utilizing a scoring system ranging from 0 to 10, where higher scores indicate worse respiratory status. The analysis will focus on the sensitivity and specificity of individual sonographic components, with OLD diagnosis as the outcome variable.
Impact of Smoking Status on Sonographic Scoring Accuracy for OLD | 12 Months
  This analysis will measure the effect of smoking status on the diagnostic accuracy of the sonographic score for OLD, employing a scoring system from 0 to 10, where higher scores reflect worse respiratory health. Using regression analysis, the outcome will include estimates of the impact of smoking status on the probability of OLD diagnosis, adjusting for the sonographic score, and will quantify the additional diagnostic value provided by smoking status information.

CONTACTS AND LOCATIONS:
Overall Officials: Lior Fuchs, MD, Principal Investigator — Soroka University Medical Center
Locations (1):
- Soroka University Medical Center, Beersheba, South, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moore CL, Copel JA. Point-of-care ultrasonography. N Engl J Med. 2011 Feb 24;364(8):749-57. doi: 10.1056/NEJMra0909487. No abstract available. PMID 21345104
- [Background] Mayo PH, Copetti R, Feller-Kopman D, Mathis G, Maury E, Mongodi S, Mojoli F, Volpicelli G, Zanobetti M. Thoracic ultrasonography: a narrative review. Intensive Care Med. 2019 Sep;45(9):1200-1211. doi: 10.1007/s00134-019-05725-8. Epub 2019 Aug 15. PMID 31418060
- [Background] Johri AM, Durbin J, Newbigging J, Tanzola R, Chow R, De S, Tam J. Cardiac Point-of-Care Ultrasound: State-of-the-Art in Medical School Education. J Am Soc Echocardiogr. 2018 Jul;31(7):749-760. doi: 10.1016/j.echo.2018.01.014. Epub 2018 Mar 15. PMID 29550326
- [Background] Sekiguchi H. Tools of the Trade: Point-of-Care Ultrasonography as a Stethoscope. Semin Respir Crit Care Med. 2016 Feb;37(1):68-87. doi: 10.1055/s-0035-1570353. Epub 2016 Feb 4. PMID 26844609
- [Background] Alrajab S, Youssef AM, Akkus NI, Caldito G. Pleural ultrasonography versus chest radiography for the diagnosis of pneumothorax: review of the literature and meta-analysis. Crit Care. 2013 Sep 23;17(5):R208. doi: 10.1186/cc13016. PMID 24060427
- [Background] Shah VP, Tunik MG, Tsung JW. Prospective evaluation of point-of-care ultrasonography for the diagnosis of pneumonia in children and young adults. JAMA Pediatr. 2013 Feb;167(2):119-25. doi: 10.1001/2013.jamapediatrics.107. PMID 23229753
- [Background] Nazerian P, Vanni S, Volpicelli G, Gigli C, Zanobetti M, Bartolucci M, Ciavattone A, Lamorte A, Veltri A, Fabbri A, Grifoni S. Accuracy of point-of-care multiorgan ultrasonography for the diagnosis of pulmonary embolism. Chest. 2014 May;145(5):950-957. doi: 10.1378/chest.13-1087. PMID 24092475
- [Background] Diaz-Gomez JL, Mayo PH, Koenig SJ. Point-of-Care Ultrasonography. N Engl J Med. 2021 Oct 21;385(17):1593-1602. doi: 10.1056/NEJMra1916062. No abstract available. PMID 34670045
- [Background] Qaseem A, Etxeandia-Ikobaltzeta I, Mustafa RA, Kansagara D, Fitterman N, Wilt TJ; Clinical Guidelines Committee of the American College of Physicians; Batur P, Cooney TG, Crandall CJ, Hicks LA, Lin JS, Maroto M, Tice J, Tufte JE, Vijan S, Williams JW Jr. Appropriate Use of Point-of-Care Ultrasonography in Patients With Acute Dyspnea in Emergency Department or Inpatient Settings: A Clinical Guideline From the American College of Physicians. Ann Intern Med. 2021 Jul;174(7):985-993. doi: 10.7326/M20-7844. Epub 2021 Apr 27. PMID 33900792
- [Background] Zanobetti M, Scorpiniti M, Gigli C, Nazerian P, Vanni S, Innocenti F, Stefanone VT, Savinelli C, Coppa A, Bigiarini S, Caldi F, Tassinari I, Conti A, Grifoni S, Pini R. Point-of-Care Ultrasonography for Evaluation of Acute Dyspnea in the ED. Chest. 2017 Jun;151(6):1295-1301. doi: 10.1016/j.chest.2017.02.003. Epub 2017 Feb 16. PMID 28212836
- [Background] Lichtenstein DA, Meziere GA. Relevance of lung ultrasound in the diagnosis of acute respiratory failure: the BLUE protocol. Chest. 2008 Jul;134(1):117-25. doi: 10.1378/chest.07-2800. Epub 2008 Apr 10. PMID 18403664
- [Background] Szalontai K, Gemes N, Furak J, Varga T, Neuperger P, Balog JA, Puskas LG, Szebeni GJ. Chronic Obstructive Pulmonary Disease: Epidemiology, Biomarkers, and Paving the Way to Lung Cancer. J Clin Med. 2021 Jun 29;10(13):2889. doi: 10.3390/jcm10132889. PMID 34209651

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT06251271/Prot_SAP_001.pdf